CLINICAL TRIAL: NCT05298254
Title: A Phase I/II, Observer-blind, Randomised, Placebo-controlled, Multi-country Study to Evaluate Reactogenicity, Safety, Immune Response, and Efficacy of an HSV-targeted Immunotherapy in Healthy Participants Aged 18-40 Years or in Participants Aged 18-60 Years With Recurrent Genital Herpes
Brief Title: A Study on the Reactogenicity, Safety, Immune Response, and Efficacy of a Targeted Immunotherapy Against HSV in Healthy Participants Aged 18-40 Years or in Participants Aged 18-60 Years With Recurrent Genital Herpes
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 215336; 2021-003586-35 (EudraCT Number)
Record Dates: First submitted 2022-03-04; First posted 2022-03-28 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Herpes Simplex
Keywords: First Time in Human; Healthy participants; Recurrent genital herpes; Herpes Simplex Virus; Reactogenicity; Safety; Immune response; Efficacy
MeSH Terms: conditions — Herpes Simplex; Herpes Genitalis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Data will be collected in an observer-blind manner.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (13):
- Non-adjuvanted HSV formulation 1 - Part I Group (Experimental): Participants enrolled in Part I of the study who receive 2 doses of the non-adjuvanted HSV formulation 1 vaccine, one at Day 1 and one at Day 29.
  Interventions: Biological: Non-adjuvanted HSV formulation 1
- Non-adjuvanted HSV formulation 2 - Part I Group (Experimental): Participants enrolled in Part I of the study who receive 2 doses of the non-adjuvanted HSV formulation 2 vaccine, one at Day 1 and one at Day 29.
  Interventions: Biological: Non-adjuvanted HSV formulation 2
- Non-adjuvanted HSV formulation 3 - Part I Group (Experimental): Participants enrolled in Part I of the study who receive 2 doses of the non-adjuvanted HSV formulation 3 vaccine, one at Day 1 and one at Day 29.
  Interventions: Biological: Non-adjuvanted HSV formulation 3
- HSV formulation 1 with adjuvant 1 - Part I Group (Experimental): Participants enrolled in Part I of the study who receive 2 doses of the HSV formulation 1 with adjuvant 1 vaccine, one at Day 1 and one at Day 29.
  Interventions: Biological: HSV formulation 1 with adjuvant 1
- HSV formulation 2 with adjuvant 1 - Part I Group (Experimental): Participants enrolled in Part I of the study who receive 2 doses of the HSV formulation 2 with adjuvant 1 vaccine, one at Day 1 and one at Day 29.
  Interventions: Biological: HSV formulation 2 with adjuvant 1
- HSV formulation 3 with adjuvant 1 - Part I Group (Experimental): Participants enrolled in Part I of the study who receive 2 doses of the HSV formulation 3 with adjuvant 1 vaccine, one at Day 1 and one at Day 29.
  Interventions: Biological: HSV formulation 3 with adjuvant 1
- HSV formulation 1 with adjuvant 2 - Part I Group (Experimental): Participants enrolled in Part I of the study who receive 2 doses of the HSV formulation 1 with adjuvant 2 vaccine, one at Day 1 and one at Day 29.
  Interventions: Biological: HSV formulation 1 with adjuvant 2
- HSV formulation 2 with adjuvant 2 - Part I Group (Experimental): Participants enrolled in Part I of the study who receive 2 doses of the HSV formulation 2 with adjuvant 2 vaccine, one at Day 1 and one at Day 29.
  Interventions: Biological: HSV formulation 2 with adjuvant 2
- HSV formulation 3 with adjuvant 2 - Part I Group (Experimental): Participants enrolled in Part I of the study who receive 2 doses of the HSV formulation 3 with adjuvant 2 vaccine, one at Day 1 and one at Day 29.
  Interventions: Biological: HSV formulation 3 with adjuvant 2
- Placebo - Part I Group (Placebo Comparator): Participants enrolled in Part I of the study who receive 2 doses of Placebo, one at Day 1 and one at Day 29.
  Interventions: Drug: Placebo
- HSVTI formulation (F) 1 - Part II Group (Experimental): Participants enrolled in Part II of the study who receive 2 doses of the formulation of the HSVTI_F1 selected from Part I of the study, one at Day 1 and one at Day 29.
  Interventions: Biological: HSVTI_F1
- HSVTI_F2 - Part II Group (Experimental): Participants enrolled in Part II of the study who receive 2 doses of the HSVTI_F2 selected from Part I of the study, one at Day 1 and one at Day 29.
  Interventions: Biological: HSVTI_F2
- Placebo - Part II Group (Placebo Comparator): Participants enrolled in Part II of the study who receive 2 doses of Placebo, one at Day 1 and one at Day 29.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Non-adjuvanted HSV formulation 1 — Two doses of the non-adjuvanted HSV formulation 1 vaccine administered intramuscularly in the deltoid region of the non-dominant arm, one each at Day 1 and Day 29, during Part I of the study.
  Arms: Non-adjuvanted HSV formulation 1 - Part I Group
Biological: Non-adjuvanted HSV formulation 2 — Two doses of the non-adjuvanted HSV formulation 2 vaccine administered intramuscularly in the deltoid region of the non-dominant arm, one each at Day 1 and Day 29, during Part I of the study.
  Arms: Non-adjuvanted HSV formulation 2 - Part I Group
Biological: Non-adjuvanted HSV formulation 3 — Two doses of the non-adjuvanted HSV formulation 3 vaccine administered intramuscularly in the deltoid region of the non-dominant arm, one each at Day 1 and Day 29, during Part I of the study.
  Arms: Non-adjuvanted HSV formulation 3 - Part I Group
Biological: HSV formulation 1 with adjuvant 1 — Two doses of the HSV formulation 1 with adjuvant 1 vaccine administered intramuscularly in the deltoid region of the non-dominant arm, one each at Day 1 and Day 29, during Part I of the study.
  Arms: HSV formulation 1 with adjuvant 1 - Part I Group
Biological: HSV formulation 2 with adjuvant 1 — Two doses of the HSV formulation 2 with adjuvant 1 vaccine administered intramuscularly in the deltoid region of the non-dominant arm, one each at Day 1 and Day 29, during Part I of the study.
  Arms: HSV formulation 2 with adjuvant 1 - Part I Group
Biological: HSV formulation 3 with adjuvant 1 — Two doses of the HSV formulation 3 with adjuvant 1 vaccine administered intramuscularly in the deltoid region of the non-dominant arm, one each at Day 1 and Day 29, during Part I of the study.
  Arms: HSV formulation 3 with adjuvant 1 - Part I Group
Biological: HSV formulation 1 with adjuvant 2 — Two doses of the HSV formulation 1 with adjuvant 2 vaccine administered intramuscularly in the deltoid region of the non-dominant arm, one each at Day 1 and Day 29, during Part I of the study.
  Arms: HSV formulation 1 with adjuvant 2 - Part I Group
Biological: HSV formulation 2 with adjuvant 2 — Two doses of the HSV formulation 2 with adjuvant 2 vaccine administered intramuscularly in the deltoid region of the non-dominant arm, one each at Day 1 and Day 29, during Part I of the study.
  Arms: HSV formulation 2 with adjuvant 2 - Part I Group
Biological: HSV formulation 3 with adjuvant 2 — Two doses of the HSV formulation 3 with adjuvant 2 vaccine administered intramuscularly in the deltoid region of the non-dominant arm, one each at Day 1 and Day 29, during Part I of the study.
  Arms: HSV formulation 3 with adjuvant 2 - Part I Group
Drug: Placebo — Two doses of Placebo administered intramuscularly in the deltoid region of the non-dominant arm, one each at Day 1 and Day 29, during Part I and Part II of the study.
  Arms: Placebo - Part I Group; Placebo - Part II Group
Biological: HSVTI_F1 — Two doses of the formulation of the HSVTI_F1 selected from Part I of the study administered intramuscularly in the deltoid region of the non-dominant arm, one each at Day 1 and Day 29, during Part II of the study.
  Arms: HSVTI formulation (F) 1 - Part II Group
Biological: HSVTI_F2 — Two doses of the formulation of the HSVTI_F2 selected from Part I of the study administered intramuscularly in the deltoid region of the non-dominant arm, one each at Day 1 and Day 29, during Part II of the study.
  Arms: HSVTI_F2 - Part II Group

SUMMARY:
The purpose of this first-time-in-human (FTiH) study is to evaluate the reactogenicity, safety, immune response, and efficacy of an investigational herpes simplex virus (HSV)-targeted immunotherapy (TI). The study will be conducted in 2 parts: Part I assessing different formulations of the Herpes Simplex Virus-targeted immunotherapy (HSVTI) in healthy participants aged 18-40 years; Part II assessing the 2 formulations of the HSVTI in participants aged 18-60 years with recurrent genital herpes.

ELIGIBILITY:
Inclusion Criteria:

* • Participants, who, in the opinion of the investigator, can and will comply with the requirements of the Protocol.
* Written informed consent obtained from the participant prior to performance of any study-specific procedure.
* Women of non-childbearing potential can be enrolled in the study.
* Women of childbearing potential can be enrolled in the study, if the participant:

  * Has practiced highly effective contraception for one month prior to study intervention administration, and,
  * Has a negative pregnancy test result at the Screening visit and on the day of each study intervention administration, and,
  * For PART I: Has agreed to continue highly effective contraception until the end of the study.
  * For PART II: Has agreed to continue highly effective contraception until 3 months after last study intervention administration.
* Seronegative for human immunodeficiency virus (HIV), as determined by laboratory screening tests. Participants documented to be seropositive to HIV will not be eligible for study participation.
* Only for PART I: Healthy participants as established by medical history and physical examination, at the discretion of the investigator, before entering into the study.
* Only for PART I: Man or woman aged 18 to 40 years, included, at the time of the first study intervention administration.
* Only for PART I: Seronegative for HSV-2 as determined by Western blot performed at the Screening visit.
* Only for PART II: Participants with recurrent genital herpes and with no significant health problems as established by medical history and physical examination, at the discretion of the investigator, before entering the study.

  * Diagnosis of genital herpes for at least one year before the Screening visit.
  * History of self-reported or documented recurrent lesional genital herpes frequency of at least 3 and no more than 9 reported clinical recurrences in the 12 months preceding the screening visit, or, if still on suppressive therapy within 3 months before the Screening visit, prior to initiation of suppressive therapy.
* Only for PART II: Man or woman aged 18 to 60 years, included, at the time of the first study intervention administration.
* Only for PART II: Seropositive for HSV-2 as determined by serological testingperformed at the Screening visit, or having documented laboratory-confirmed HSV 2 genital herpes (i.e., HSV-2 DNA positive by a molecular technique such as polymerase chain reaction [PCR], or HSV-2 seropositive by a type-specific serology assay such as Western Blot or other immunoassay).Only for PART II (shedding sub-cohort): Participants agreeing to collect 2 swabs per day from anogenital area for the full duration of the 5 swabbing periods planned in the study.
* Only for PART II (shedding sub-cohort) after baseline completion: Participants having collected at least 45 out of 56 anogenital swabs during the baseline period.

Exclusion Criteria:

Medical Conditions

* Acute or chronic clinically significant pulmonary, cardiovascular, hepatic, endocrine, or renal functional abnormality, as determined by physical examination or laboratory screening tests.
* Any other clinical condition that, in the opinion of the investigator, might pose additional risk to the participant due to participation in the study or that would interfere with the efficacy and immunogenicity assessments planned in this study.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the study intervention.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Hypersensitivity to latex.
* Recurrent history or uncontrolled neurological disorders or seizures.
* Haematological and/or biochemical parameters outside the normal laboratory ranges at the Screening visit, unless the laboratory abnormalities are considered not clinically significant by the investigator.
* Body mass index =<18 kg/m^2 or >=35 kg/m^2.
* Past or current Guillain-Barré syndrome.
* History of any form of ocular HSV infection, HSV-related erythema multiforme, or HSV-related neurological complications.

Prior/Concomitant Therapy

* Use of any investigational or non-registered product other than the study intervention during the period beginning as of the Screening visit, or planned use during the study period.
* Planned administration/administration of a vaccine not foreseen by the Protocol in the period starting 15 days before each dose and ending 15 days after each dose of study intervention administration.
* Administration or planned administration of long-acting immune-modifying drugs at any time during the study period.
* Administration of immunoglobulins and/or any blood products or plasma derivatives during the period starting 3 months before the first dose of study intervention or planned administration during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs during the period starting 3 months prior to the first study intervention dose. For corticosteroids, this will mean prednisone equivalent >= 20 mg/day, or equivalent. Inhaled, intra articular and topical steroids are allowed.
* Prior receipt of another vaccine containing HSV antigens.
* Only for PART II: Planned use of suppressive anti-HSV therapy from the Screening visit until the end of the study.
* Only for PART II: Planned use of tenofovir therapy, or other medication known to affect HSV shedding or genital lesions from the Screening visit until the end of the study. Only for PART II: Planned use of topical antiviral medication in the anogenital region from the Screening visit until the end of the study.
* Only for PART II: Planned use of any episodic antiviral medications during the swabbing periods (including the baseline period) (only for the shedding sub-cohort).

Prior/Concurrent Clinical Study Experience

• Concurrently participating in another clinical study, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non-investigational intervention.

Other Exclusions

* Pregnant or lactating women.
* Woman planning to become pregnant or planning to discontinue contraceptive precautions in the period starting from the Screening visit up to 3 months post-last dose of study intervention.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 505 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2025-06-12 (Actual); Study Completion 2025-06-12 (Actual)

PRIMARY OUTCOMES:
Percentage of participants reporting each solicited administration site event | Within 7 days after the first study intervention dose (administered at Day 1)
  The solicited administration site events are pain, redness and swelling.
Percentage of participants reporting each solicited administration site event | Within 7 days after the second study intervention dose (administered at Day 29)
  The solicited administration site events are pain, redness and swelling.
Percentage of participants reporting each solicited systemic event | Within 7 days after the first study intervention dose (administered at Day 1)
  The solicited systemic events are fever, fatigue, headache, myalgia and arthralgia. The preferred location for measuring temperature is the oral cavity. Fever is defined as temperature equal to or above (≥) 38.0 degree Celsius (°C)/ 100.4 degree Fahrenheit (°F), regardless the location of measurement.
Percentage of participants reporting each solicited systemic event | Within 7 days after the second study intervention dose (administered at Day 29)
  The solicited systemic events are fever, fatigue, headache, myalgia and arthralgia. The preferred location for measuring temperature is the oral cavity. Fever is defined as temperature equal to or above (≥) 38.0 degree Celsius (°C)/ 100.4 degree Fahrenheit (°F), regardless the location of measurement.
Percentage of participants reporting unsolicited adverse events (AEs) | Within 28 days after the first study intervention dose (administered at Day 1)
  An unsolicited AE is any AE reported in addition to those solicited during the clinical study. Also, any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms (7 days after each dose) is reported as an unsolicited AE.
Percentage of participants reporting unsolicited adverse events (AEs) | Within 28 days after the second study intervention dose (administered at Day 29)
  An unsolicited AE is any AE reported in addition to those solicited during the clinical study. Also, any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms (7 days after each dose) is reported as an unsolicited AE.
Percentage of participants reporting medically attended events (MAEs) | From Dose 1 (Day 1) up 12 months after last study intervention administration (Day 394)
  An MAE is an unsolicited AE for which the participants received medical attention defined as any symptoms or illnesses requiring hospitalization, or an emergency room visit, or visit to/by healthcare professionals.
Percentage of participants reporting any serious adverse events (SAEs) | From Dose 1 (Day 1) up to 12 months after last study intervention administration (Day 394)
  An SAE is any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study participant or results in abnormal pregnancy outcomes.
Percentage of participants reporting any potential immune-mediated disease (pIMDs) (classified as newly diagnosed or exacerbation of pre-existing events) | From Dose 1 (Day 1) up to 12 months after last study intervention administration (Day 394)
  PIMDs are a subset of adverse events of special interest (AESIs) that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune aetiology.
Percentage of participants reporting any haematological and biochemical laboratory abnormalities at pre-study intervention administration (Day 1) in Part I of the study | At pre-study intervention administration (Day 1)
  Clinically significant haematological and biochemical abnormal laboratory findings are those which are not associated with an underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition.
Percentage of participants reporting any haematological and biochemical laboratory abnormalities at Day 8 in Part I of the study | At Day 8
Percentage of participants reporting any haematological and biochemical laboratory abnormalities at Day 29 in Part I of the study | At Day 29
Percentage of participants reporting any haematological and biochemical laboratory abnormalities at Day 36 in Part I of the study | At Day 36
Percentage of participants reporting any haematological and biochemical laboratory abnormalities at Day 64 in Part I of the study | At Day 64
Percentage of participants reporting any haematological and biochemical laboratory abnormalities at pre-study intervention administration (Day 1) in Part II of the study | At pre-study intervention administration (Day 1)
Percentage of participants reporting any haematological and biochemical laboratory abnormalities at Day 8 in Part II of the study | At Day 8
Percentage of participants reporting any haematological and biochemical laboratory abnormalities at Day 29 in part II of the study | At Day 29
Percentage of participants reporting any haematological and biochemical laboratory abnormalities at Day 36 in Part II of the study | At Day 36
Percentage of participants reporting any haematological and biochemical laboratory abnormalities at Day 57 in Part II of the study | At Day 57
Time-to-first confirmed HSV-2 RGH episode in Part II of the study | 14 days post-Dose 2 (Day 43) to end of RGH event reporting period
  A suspected RGH episode will be classified as confirmed HSV-2 RGH episode if at least one of the lesional or anogenital swabs taken during the concerned episode is positive for HSV-2 as measured by PCR. The end of RGH reporting can occur at Day 209 for participants who have not yet completed Visit 8 [Day 209] at the time the Informed Consent Form (ICF) addendum was signed and consented, or at non-scheduled time, being defined by the date on which participants decided to stop the RGH reporting after acknowledgement of unsuccessful primary analysis before ICF addendum consent or the day the eDiary is deactivated after ICF addendum consent.

SECONDARY OUTCOMES:
Number of confirmed HSV-2 RGH episodes in Part II of the study | 14 days post-Dose 2 (Day 43) to end of RGH event reporting period
  A suspected RGH episode will be classified as confirmed HSV-2 RGH episode if at least one of the lesional or anogenital swabs taken during the concerned episode is positive for HSV-2 as measured by PCR. The end of RGH reporting can occur at Day 209 for participants who have not yet completed Visit 8 [Day 209] at the time the Informed Consent Form (ICF) addendum was signed and consented, or at non-scheduled time, being defined by the date on which participants decided to stop the RGH reporting after acknowledgement of unsuccessful primary analysis before ICF addendum consent or the day the eDiary is deactivated after ICF addendum consent.
Percentage of participants free from confirmed HSV-2 RGH episode in Part II of the study | At 6 months after the last study intervention administration (Day 29)
  A suspected RGH episode will be classified as confirmed HSV-2 RGH episode if at least one of the lesional or anogenital swabs taken during the concerned episode is positive for HSV-2 as measured by PCR.
Herpes Symptoms Checklist (HSC) total score during each confirmed HSV-2 RGH episode in Part II of the study | 14 days post-Dose 2 (Day 43) to end of RGH event reporting period
  During genital herpes recurrences, participants are asked to complete the HSC, a 13-item checklist of herpes symptoms, where respondents record the severity of symptoms on a 4-point scale where 0 indicates no symptom and a higher point for more symptoms and severity. Total scores range from 0 (no symptom) to 39 (severe symptoms). At the onset of the genital herpes recurrence, this questionnaire is to be completed once daily, until no lesions or symptoms are present. The end of RGH reporting can occur at Day 209 for participants who have not yet completed Visit 8 [Day 209] at the time the Informed Consent Form (ICF) addendum was signed and consented, or at non-scheduled time, being defined by the date on which participants decided to stop the RGH reporting after acknowledgement of unsuccessful primary analysis before ICF addendum consent or the day the eDiary is deactivated after ICF addendum consent.
Number of days with RGH-associated symptoms during each confirmed HSV-2 RGH episode in Part II of the study | 14 days post-Dose 2 (Day 43) to end of RGH event reporting period
  Duration in days (i.e., number of days with RGH-associated symptoms) of each genital herpes recurrence is displayed by arm group. The end of RGH reporting can occur at Day 209 for participants who have not yet completed Visit 8 [Day 209] at the time the Informed Consent Form (ICF) addendum was signed and consented, or at non-scheduled time, being defined by the date on which participants decided to stop the RGH reporting after acknowledgement of unsuccessful primary analysis before ICF addendum consent or the day the eDiary is deactivated after ICF addendum consent.
Number of days with confirmed HSV-2 genital herpes lesions in Part II of the study | 14 days post-Dose 2 (Day 43) to end of RGH event reporting period
  Number of days on which lesions (swelling, blisters, sores, or crusts) are reported by the participant in the anogenital area during confirmed RGH episodes divided by the number of days of follow-up. The end of RGH reporting can occur at Day 209 for participants who have not yet completed Visit 8 [Day 209] at the time the Informed Consent Form (ICF) addendum was signed and consented, or at non-scheduled time, being defined by the date on which participants decided to stop the RGH reporting after acknowledgement of unsuccessful primary analysis before ICF addendum consent or the day the eDiary is deactivated after ICF addendum consent.
HSV-2 shedding rate reduction from baseline to 6 weeks post-Dose 2 (Day 71) in Part II of the study | At 6 weeks post-Dose 2 (Day 71) compared to baseline (Day -28 to Day -1)
  The HSV-2 shedding rate reduction is calculated as 1- (the HSV-2 shedding rate one month post-Dose 2 divided by the baseline HSV-2 shedding rate)*100.
Number of HSV-2 DNA shedding episodes in Part II of the study | Day -28 to Day -1
  Number of HSV-2 shedding episodes during the 28-day swabbing period.
Number of HSV-2 DNA shedding episodes in Part II of the study | Day 43 to Day 70
  Number of HSV-2 shedding episodes during the 28-day swabbing period.
Number of HSV-2 DNA shedding episodes in Part II of the study | Day 181 to Day 208
  Number of HSV-2 shedding episodes during the 28-day swabbing period.
Duration of HSV-2 DNA shedding episodes in Part II of the study | Day -28 to Day -1
  Number of days of a HSV-2 shedding episode.
Duration of HSV-2 DNA shedding episodes in Part II of the study | Day 43 to Day 70
  Number of days of a HSV-2 shedding episode.
Duration of HSV-2 DNA shedding episodes in Part II of the study | Day 181 to Day 208
  Number of days of a HSV-2 shedding episode.
Anti-HSVTI antibody geometric mean concentrations (GMCs) in Part I of the study | At pre-study intervention administration (Day 1), Day 29, Day 64, Day 209 and Day 394
Anti-HSVTI antibody geometric mean concentrations (GMCs) in Part II of the study | At pre-study intervention administration (Day 1), Day 29 and Day 57
Percentage of seropositive participants for anti-HSVTI antibodies in Part I of the study | At pre-study intervention administration (Day 1), Day 29, Day 64, Day 209 and Day 394
Percentage of seropositive participants for anti-HSVTI antibodies in Part II of the study | At pre-study intervention administration (Day 1), Day 29 and Day 57
Geometric mean of HSVTI-specific Cluster of Differentiation (CD)4+ T-cells frequency expressing at least two activation markers and including at least one cytokine in Part I of the study | At pre-study intervention administration (Day 1), Day 29, Day 64, Day 209 and Day 394
Geometric mean of HSVTI-specific CD4+ T-cells frequency expressing at least 2 activation markers and including at least 1 cytokine in Part II of the study | At pre-study intervention administration (Day 1), Day 29 and Day 57
Geometric mean of HSVTI-specific CD8+ T-cells frequency expressing at least two activation markers and including at least one cytokine in Part I of the study | At pre-study intervention administration (Day 1), Day 29, Day 64, Day 209 and Day 394
Geometric mean of HSVTI-specific CD8+ T-cells frequency expressing at least 2 activation markers and including at least 1 cytokine in Part II of the study | At pre-study intervention administration (Day 1), Day 29 and Day 57

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (26):
- United States (6):
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Seattle, Washington
- Australia (2):
  - GSK Investigational Site, Darlinghurst, New South Wales
  - GSK Investigational Site, Sydney, New South Wales
- Belgium (4):
  - GSK Investigational Site, Antwerp
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Edegem
  - GSK Investigational Site, Ghent
- GSK Investigational Site, Montreal, Quebec, Canada
- GSK Investigational Site, Tartu, Estonia
- Germany (5):
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Bochum
  - GSK Investigational Site, Cologne
  - GSK Investigational Site, Frankfurt
  - GSK Investigational Site, Hamburg
- Spain (3):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Marbella
- United Kingdom (4):
  - GSK Investigational Site, Brighton
  - GSK Investigational Site, Liverpool
  - GSK Investigational Site, London
  - GSK Investigational Site, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Study Sponsor will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gskstudyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, a key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.gskstudyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf